CLINICAL TRIAL: NCT03131388
Title: Clinical Performance Evaluation of AMH Assay
Status: Completed | Type: Observational
Sponsor: Beckman Coulter, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AMH 2.7.1
Record Dates: First submitted 2017-04-17; First posted 2017-04-27 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Anti-Mullerian Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Access AMH Assay

SUMMARY:
The Access AMH Assay is an in vitro diagnostic assay intended as an aid for fertility assessment. The purpose of the study is to evaluate the clinical performance of the Access AMH Assay in the intended use population.

DETAILED DESCRIPTION:
same as brief summary

ELIGIBILITY:
Inclusion Criteria:

* ≥ 21 and < 46 years of age
* Regular menstrual cycle
* Both ovaries present

Exclusion Criteria:

* Evidence of PCOS
* Confirmed ovarian endometrioma
* Ovarian surgery prior to enrollment
* Being treated for cancer
* Hormonal contraceptive use prior to enrollment
* Currently pregnant

Ages: 21 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Adult women presenting to fertility clinics for fertility assessment
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Measurement of AMH as an aid for fertility assessment | Day 2 to 4 of menstrual cycle
  Comparison of AMH levels in women at different levels of AFC to aid in assessing ovarian reserve

CONTACTS AND LOCATIONS:
Overall Officials: Fred Siebert, Study Director — Beckman Coulter
Locations (13):
- United States (12):
  - BRI, Phoenix, Arizona
  - Stanford, Palo Alto, California
  - FSMG, San Diego, California
  - RAD, Newark, Delaware
  - WRMG, Clearwater, Florida
  - Vios Fertility, Swansea, Illinois
  - BIVF, Waltham, Massachusetts
  - Mainline Fertility, Bryn Mawr, Pennsylvania
  - Univ Pennsylvania, Philadelphia, Pennsylvania
  - CARE, Dallas, Texas
  - CORM, Webster, Texas
  - PNWF, Seattle, Washington
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No